CLINICAL TRIAL: NCT03339947
Title: Poor Knowledge Among French Travelers of the Risk of Acquiring Multidrug-resistant Bacteria During Travel
Brief Title: French Travelers' Knowledge of Risk of Acquiring ESBL-PE
Acronym: MDR bacteria
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2016Ao006
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Travel Medicine
Keywords: Multidrug-resistant Enterobacteriaceae acquisition; travellers' diarrhoea; international travel
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Travel medicine: All adult travellers who attended the consultation for travel medicine and international vaccination in Reims University Hospital.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
Since it is not routine practice in France to raise public awareness about the risk of acquiring multidrug resistant Enterobacteriaceae (MRE) during international travel, the investigators aimed to determine, among French travelers attending a consultation for travel medicine, patients level of knowledge about the risk of acquiring MRE.

DETAILED DESCRIPTION:
Since it is not routine practice in France to raise public awareness about the risk of acquiring multidrug resistant Enterobacteriaceae (MRE) during international travel, The investigators aimed to assess, among persons attending a consultation for travel medicine and international vaccines, patients level of knowledge regarding the risk of acquiring MRE, preventive behaviours and the need to inform health professionals that they had recently travelled if the patients require medical care after their return. A cross-sectional study was performed in the consultation for travel medicine and international vaccination in Reims University Hospital, France. All adult travellers who attended this consultation between January 2016 and May 2016 and who completed the questionnaire were included in the study. The questionnaire was completed before the planned travel. The travellers answered the questionnaires before seeing the physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult travellers who attended the consultation for travel medicine and international vaccination in Reims University Hospital
* Adult who completed the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult travellers who attended the consultation for travel medicine and international vaccination in Reims University Hospital between January 2016 and May 2016 and who completed the questionnaire were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Level of knowledge regarding multidrug resistant Enterobacteriaceae | Day 1
  The questionnaire was completed before the planned travel and recorded information on the patient's knowledge of the definition of multidrug resistant bacteria (MDR), knowledge of the factors associated with acquiring MDR bacteria, consumption of antibiotics during previous travel, awareness of the need to inform health professionals about the recent trip in case of health problems after return, perceived need for more information about MDR bacteria, desired source of such information. The questions about knowledge were designed to be as simple as possible, with closed answers ('yes', 'no', 'don't know')

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Migault C, Kanagaratnam L, Nguyen Y, Lebrun D, Giltat A, Hentzien M, Bajolet O, Drame M, Bani-Sadr F. Poor knowledge among French travellers of the risk of acquiring multidrug-resistant bacteria during travel. J Travel Med. 2016 Oct 30;24(1):taw073. doi: 10.1093/jtm/taw073. Print 2016 Jul. No abstract available. PMID 27799500